CLINICAL TRIAL: NCT02216552
Title: Safety and Efficacy of Resveratrol for the Treatment of Non-Alcoholic Fatty Liver Disease and Associated Insulin Resistance in Overweight and Obese Adolescents
Brief Title: Resveratrol for the Treatment of Non Alcoholic Fatty Liver Disease and Insulin Resistance in Overweight Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Brandy Wicklow, Principal Investigator MD, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013-01-15-RESV
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: NAFLD; TYPE 2 DIABETES; METABOLIC SYNDROME
Keywords: Pediatrics; Adolescents; NAFLD; Spectroscopy; Type 2 diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: Resveratrol as ResVida (TM) compared to a placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Experimental): Intervention: Resveratrol Oral supplementation of resveratrol (ResVida) 75 mg twice daily (with breakfast and dinner) for a total daily dose of 150 mg for the duration of 30 days.
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Intervention: Placebo Control Oral supplementation of placebo twice daily (with breakfast and dinner) for a total duration of 30 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — All adolescents will receive standardized lifestyle counselling at enrolment designed and disseminated by a registered dietitian as well as a licensed physiotherapist who both have experience working with overweight adolescents. The lifestyle component will be goal-based and tailored to each participant. The overall content and messaging will be consistent for all participants with nutritional recommendations based on Canada Food Guide and physical activity counselling aligning with the Healthy Active Living Recommendations of the Canadian Pediatric Society and Health Canada's Physical Activity Guidelines.
  Other Names: ResVida (Registered Trademark of DSM)
  Arms: Resveratrol
Dietary Supplement: Placebo — All adolescents will receive standardized lifestyle counselling at enrolment designed and disseminated by a registered dietitian as well as a licensed physiotherapist who both have experience working with overweight adolescents. The lifestyle component will be goal-based and tailored to each participant. The overall content and messaging will be consistent for all participants with nutritional recommendations based on Canada Food Guide and physical activity counselling aligning with the Healthy Active Living Recommendations of the Canadian Pediatric Society and Health Canada's Physical Activity Guidelines.
  Arms: Placebo

SUMMARY:
The current project is designed as a 30-day pilot trial to demonstrate the safety and tolerability of resveratrol therapy in overweight adolescents to decrease liver fat, and improve insulin sensitivity to prevent type 2 diabetes.

DETAILED DESCRIPTION:
Pilot study of 10 overweight or obese children with MRS determined fatty liver randomized to resveratrol or placebo. Primary outcome measures include change in liver triglyceride content as determined by MRS and improvement in insulin resistance as determined by the area under the curve of glucose excursion during a 75 gram oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* 13 to <18 years of age
* BMI considered overweight (BMI > 25 kg/m2 ) or obese (BMI > 30 kg/m2 )
* Confirmed 1H-MRS defined hepatic steatosis (>5.5% fat/water)
* Parent/Guardian willing and able to provide written, signed informed consent, and subjects willing to co-sign parental consent
* Sexually active subjects must be willing to use an acceptable method of contraception
* Females of child bearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* The use of any chronic medications with the exception of oral birth control and natural health products with the exception of multivitamins.
* Adolescents with altered insulin sensitivity or tissue lipid content unrelated to obesity and the metabolic syndrome, including:

type 2 diabetes; present or previous malignancy renal disease, hypertension (anyone who has BPs over the 99th percentile for age and gender) or liver disease;

* significant weight loss (10% in last six months) or enrolled in weight loss program in the six months prior to the study;
* self-reported history of alcohol consumption of greater than two drinks per day and/or drinking alcohol more than once weekly;
* report using non-prescription recreational drugs;
* allergies or sensitivities to any of the ingredients in the investigational product or placebo;
* females breastfeeding at screening or planning on becoming pregnant at any time during the study;

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01-01 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Safety/ Adverse Event Outcome | One week
  1. Primary Side effect profile determined by participant interview and serum biochemistry. Side effect profile determined by serum biochemistry: AST, ALT, total and conjugated bilirubin, Creatinine, sodium, potassium, calcium, magnesium, chloride and TC02, haemoglobin, haematocrit, white blood cell and platelet counts, erythrocytes, and fasting lipid levels (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides). Fasting glucose and insulin levels. PT/INR and PTT levels.
  2. Vital signs
Safety/ Adverse Event Outcome | Week 2
  1. Primary Side effect profile determined by participant interview. Side effect profile determined by serum biochemistry: AST, ALT, total and conjugated bilirubin, Creatinine, sodium, potassium, calcium, magnesium, chloride and TC02, haemoglobin, haematocrit, white blood cell and platelet counts, erythrocytes, and fasting lipid levels (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides). Fasting glucose and insulin levels. PT/INR and PTT levels.
  2. Vital signs
Safety/ Adverse Event Outcome | Week 3
  1. Primary Side effect profile determined by participant interview. Side effect profile determined by serum biochemistry: AST, ALT, total and conjugated bilirubin, Creatinine, sodium, potassium, calcium, magnesium, chloride and TC02, haemoglobin, haematocrit, white blood cell and platelet counts, erythrocytes, and fasting lipid levels (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides). Fasting glucose and insulin levels. PT/INR and PTT levels.
  2. Vital signs
Safety/ Adverse Event Outcome | Week 4
  1. Primary Side effect profile determined by participant interview. Side effect profile determined by serum biochemistry: AST, ALT, total and conjugated bilirubin, Creatinine, sodium, potassium, calcium, magnesium, chloride and TC02, haemoglobin, haematocrit, white blood cell and platelet counts, erythrocytes, and fasting lipid levels (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides). Fasting glucose and insulin levels. PT/INR and PTT levels.
  2. Vital signs
Safety/ Adverse Event Outcome | Week 8
  1. Primary Side effect profile determined by participant interview. Side effect profile determined by serum biochemistry: AST, ALT, total and conjugated bilirubin, Creatinine, sodium, potassium, calcium, magnesium, chloride and TC02, haemoglobin, haematocrit, white blood cell and platelet counts, erythrocytes, and fasting lipid levels (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides). Fasting glucose and insulin levels. PT/INR and PTT levels.
  2. Vital signs
Efficacy Outcome | Week 4
  To determine efficacy of resveratrol to reduce hepatic and cardiac triglyceride content in adolescents with NAFL MR spectroscopy will be performed using a 3.0-Tesla whole-body magnet. Sixty-four spectra will be acquired and averaged for the determination of intracellular water and lipid content. LCModel software will be used to isolate and quantify lipid and water peaks. Hepatic steatosis will be defined as hepatic triglyceride content of >.5% fat/water.

SECONDARY OUTCOMES:
Efficacy Outcome | Week 4
  To determine efficacy of resveratrol to reduce whole body insulin resistance in overweight and obese adolescents with NAFL. The 3-hr frequently sampled oral glucose tolerance test (OGTT) using a standard 75-gram-glucose-load will be performed at the baseline visit and after completion of supplementation (day 30; visit 3). Blood samples will be collected at 20, 30, 60, 90, 120 and 180 minutes after ingestion of glucose will be used for the determination of insulin sensitivity using the Matsuda index
Efficacy Outcome | Week 4
  To determine the effects of resveratrol on cardiac function and morphology in the study population. Cardiac function and morphology will be measured using a cardiac ultrasound at baseline (day 0) and at completion of supplementation (day 30; visit 3).
Efficacy Outcome | Week 1
  To determine the effect of resveratrol supplementation on serum markers of inflammation. Inflammatory markers will be assessed by measurements of circulating adiponectin, leptin, CRP, ESR, TNFalpha, IL-1beta, IL-6, and IL-10, using commercially available ELISA assays.
Efficacy Outcome | Week 2
  To determine the effect of resveratrol supplementation on serum markers of inflammation. Inflammatory markers will be assessed by measurements of circulating adiponectin, leptin, CRP, ESR, TNFalpha, IL-1beta, IL-6, and IL-10, using commercially available ELISA assays.
Efficacy Outcome | Week 3
  To determine the effect of resveratrol supplementation on serum markers of inflammation. Inflammatory markers will be assessed by measurements of circulating adiponectin, leptin, CRP, ESR, TNFalpha, IL-1beta, IL-6, and IL-10, using commercially available ELISA assays
Efficacy Outcome | Week 4
  To determine the effect of resveratrol supplementation on serum markers of inflammation. Inflammatory markers will be assessed by measurements of circulating adiponectin, leptin, CRP, ESR, TNFalpha, IL-1beta, IL-6, and IL-10, using commercially available ELISA assays

CONTACTS AND LOCATIONS:
Overall Officials: Brandy A Wicklow, MD, MSc, Principal Investigator — University of Manitoba
Locations (1):
- Children's Hospital Research Institute of Manitoba/University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No